CLINICAL TRIAL: NCT03711773
Title: Outcomes of Low-Impact Group Exercise Program for People With Ankle, Knee, and/or Hip Pain
Brief Title: Outcomes of Low-Impact Exercise Program for People With Ankle, Knee, and/or Hip Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, James Cook, Professor, Orthopedic Surgery, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012532
Record Dates: First submitted 2018-10-16; First posted 2018-10-18 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis; Osteoarthritis, Knee; Osteoarthritis, Hip; Osteoarthritis Ankle
Keywords: joint pain; osteoarthritis; hip pain; knee pain; ankle pain
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Osteoarthritis, Hip; Arthralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group Physical Therapy Class (Experimental): Group Physical Therapy Classes. Three times weekly, these subjects will have one hour group physical therapy sessions with either a physical therapist, physical therapy assistant, or personal trainer. These sessions will be aimed to improve strength and function in a low-impact setting designed specifically for those with joint pain.
  Interventions: Other: Group Physical Therapy Classes

INTERVENTIONS:
Other: Group Physical Therapy Classes — Three times weekly, these subjects will have one hour group physical therapy sessions with either a physical therapist, physical therapy assistant, or personal trainer. These sessions will be aimed to improve strength and function in a low-impact setting designed specifically for those with joint pain.

SUMMARY:
The primary objective of this study is to study how low-impact group exercise classes affect pain scores in patients with knee, hip, and ankle pain when paired with concurrent standard of care dietitian and behavioral health consults.

DETAILED DESCRIPTION:
Osteoarthritis is estimated to affect at least 10% of men and 13% of women over 60 years old in the United States. It's estimated roughly 1 million total joint replacements are being performed each year. Studies have suggested that for patients with knee pain that have high BMIs, low strength, and/or have not participated in conservative measures, a low-impact exercise plan when paired with diet counseling and behavioral health classes can improve patient reported outcomes scores in both pain and function. This study seeks to build upon this research and will provide low-impact exercise plans that will be paired with standard of care dietician and behavioral health interventions in order to offer patients a full-scope approach to battling osteoarthritis pain, especially for those with high BMIs, low strength, and/or for patients that have not attempted conservative therapy in the past. We will include patients with knee, hip, and ankle pain.

ELIGIBILITY:
Inclusion Criteria:

* 18 and over
* Ability to attend classes 3x weekly for 6 months with at least a 66% attendance rate
* Ability to concurrently attend standard of care dietitian and behavioral health classes for 6 months
* Joint pain (knee, ankle, hip)

Exclusion Criteria:

* Pregnant
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
VAS Pain scores | 6 Months
  Subjects will receive VAS pain surveys each group therapy class. These VAS pain scores (visual analog survey) are taken rated between 0, which is no pain, and 10, which is the most pain.

SECONDARY OUTCOMES:
BMI | 6 Months
  Subjects will have routine weight measurements and BMI will be calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Missouri Orthopaedic Institute, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No